CLINICAL TRIAL: NCT06316440
Title: Effect of Noise Isolation During General Anesthesia on the Incidence of Moderate to Severe Postoperative Pain in Patients Undergoing Major Abdominal Surgery
Brief Title: Effect of Noise Isolation on the Incidence of Moderate to Severe Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Shapingba People's Hospital of Chongqing University (Unknown); The 3rd. Affiliated Hospital of Chongqing Medical University (Unknown); Chongqing Hechuan District People's Hospital (Unknown); Chongqing Qijiang District People's Hospital (Unknown); ChongGang General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: noise and postoperative pain
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain
Keywords: noise Isolation; major abdominal surgery; postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into intervention group（noise blocking） and control group（No noise blocking）
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noise-canceling Group (Experimental): Intraoperative intervention with noise-canceling earphones was performed to isolate the noise
  Interventions: Device: Wear noise-cancelling earphones
- Control Group (No Intervention): After general anesthesia, the intervention of wearing noise-canceling earphones was not given

INTERVENTIONS:
Device: Wear noise-cancelling earphones — Intervention of wearing noise-canceling earphones after general anesthesia
  Arms: Noise-canceling Group

SUMMARY:
To investigate the effect of noise isolation during general anesthesia on the incidence of moderate to severe postoperative pain in patients undergoing major abdominal surgery. The aim of this study was to determine whether noise isolation can reduce the Incidence of moderate to severe postoperative pain and analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70, both male and female.
* American Society of Anesthesiologists Classification 1-3
* Patients undergoing elective major abdominal surgery under general anesthesia(Surgery time ≥ 2h)
* Voluntarily accept patient controlled intravenous analgesia and signed informed consent

Exclusion Criteria:

* Patients with previous severe disease
* Patients with hearing abnormalities
* Patients requiring mechanical ventilation or undergoing epidural catheters or other types of regional anesthesia after surgery
* Patients with chronic preoperative pain and/or long-term analgesic use
* Patients who could not cooperate with the study for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of moderate to severe postoperative pain | From ending of the surgery to 24 hours postoperatively
  Moderate to severe postoperative pain：NRS score ≥ 4 (Pain was assessed using NRS scale of 0-10, with 0 being no pain and 10 being most painful)

SECONDARY OUTCOMES:
Patient controlled analgesia pump analgesic consumption | From the time when the surgery was completed until to 24 hours after surgery
  Analgesic requirements was assessed by recording the volume of patient controlled analgesia pump
Patient controlled analgesia pump analgesic consumption | From the time when the surgery was completed until to 48 hours after surgery
  Analgesic requirements was assessed by recording the volume of patient controlled analgesia pump
The incidence of additional analgesic requirements | From the time when the surgery was completed until to 48 hours after surgery
  the percentage of patients who received additional analgesic out of the total number of patients in the group
Maximum pain score (NRS score) at 0-48 hours postoperatively | From ending of the surgery to 48 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
The incidence of moderate to severe postoperative pain | From ending of the surgery to 48 hours postoperatively
  Moderate to severe postoperative pain：NRS score ≥ 4 (Pain was assessed using NRS scale of 0-10, with 0 being no pain and 10 being most painful)
Accumulative postoperative pain NRS | From ending of the surgery to 48 hours postoperatively
  Accumulative NRS score (Pain was assessed using NRS scale of 0-10, with 0 being no pain and 10 being most painful) at 6, 12, 24 and 48 hours after surgery

OTHER OUTCOMES:
Pain score (NRS score) at 0-6 hours postoperatively | From ending of the surgery to 6 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 6-12 hours postoperatively | From ending of the surgery to 12 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 12-24 hours postoperatively | From 12 hours postoperatively to 24 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS score) at 24-48 hours postoperatively | From 24 hours postoperatively to 48 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful

CONTACTS AND LOCATIONS:
Overall Officials: Guangyou Duan, Doctor, Study Chair — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Five years after the study